CLINICAL TRIAL: NCT03533686
Title: Comparative Study of Non-invasive Adhear Bone Conduction System to Traditional Bone Conduction Hearing Devices
Brief Title: Adhear Bone Conduction System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: University of Miami (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Principal Investigator, Hillary A Snapp, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20161220
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Unilateral

STUDY DESIGN:
Intervention Model Description: Participants who are enrolled in Aims 3 are part of a cross-over design. Participants in this group will be randomly assigned to either standard of care followed by Adhear, or Adhear followed by standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Single-Sided Deafness Adult (Aim1) Group (Experimental): Adult participants with single-sided deafness and are experienced bone conduction device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant will be provided with the Adhear system for 2 weeks (plus up to 90 days).
  Interventions: Device: Adhear Bone Conduction System
- Conductive Hearing Loss Adult (Aim 2) Group (Experimental): Adult participants with conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant will be provided with the Adhear system for 2 weeks (plus up to 90 days).
  Interventions: Device: Adhear Bone Conduction System
- Adhear followed by BAHA (Aim 3) Group (Experimental): Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss or single-sided deafness who have not previously used a bone conduction device, will be provided with the Adhear system for 3 weeks (plus up to 90 days) followed by bone anchored hearing aid (BAHA) for another 3 weeks (plus up to 90 days).
  Interventions: Device: Adhear Bone Conduction System; Device: Bone anchored hearing aid (BAHA)
- BAHA followed by Adhear (Aim 3) Group (Experimental): Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss or single-sided deafness who have not previously used a bone conduction device, will be provided with the BAHA system for 3 weeks (plus up to 90 days) followed by Adhear for another 3 weeks (plus up to 90 days).
  Interventions: Device: Adhear Bone Conduction System; Device: Bone anchored hearing aid (BAHA)
- Pediatric Unilateral Conductive Hearing Loss (Aim 3a) Group (Experimental): Pediatric participants (aged 2-17 years) and their parents with unilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system for 2 weeks (plus up to 90 days).
  Interventions: Device: Adhear Bone Conduction System
- Pediatric Bilateral Conductive Hearing Loss (Aim 3b) Group (Experimental): Pediatric participants (aged 2-17 years) and their parents with bilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system. Participants who are fitted bilaterally will receive 2 Adhear systems (one for each ear) for 2 weeks (plus up to 90 days) at Visit 1. Participants who are fitted unilaterally will receive 1 Adhear system for 2 weeks (plus up to 90 days) at Visit 1, afterwards, will be fitted bilaterally at Visit 2 and receive the Adhear system for both ears for another 2 weeks (plus up to 90 days) for a total of 4 weeks (plus up to 180 days).
  Interventions: Device: Adhear Bone Conduction System

INTERVENTIONS:
Device: Adhear Bone Conduction System — Non-invasive bone conduction hearing device using adhesive
Device: Bone anchored hearing aid (BAHA) — Non-invasive bone conduction hearing device using a headband
  Arms: Adhear followed by BAHA (Aim 3) Group; BAHA followed by Adhear (Aim 3) Group

SUMMARY:
The purpose of this research study is to learn about the hearing outcomes of adult and pediatric patients who are treated with or are candidates for bone conductive devices (also termed "BAHA"). Hearing outcomes will also be assessed with a second audio processor device called the Adhear System.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2:

* Adult English speaking patients who are experienced users of Bone Anchored Implants (BAIs) for the indication of either single sided deafness or conductive hearing loss.
* Experienced will be defined as greater than 6 months of device use and no intermittent function of the device within 2 weeks of enrollment.
* Subjects will be limited to those who have normal hearing by bone conduction defined as a pure tone average of 25 dBHL or better at 500, 1000, 2000, & 3000 Hz in at least one ear.

Aim 3:

* English speaking children 5 to 17 years of age and their primary guardian who present to the clinic for treatment by BAI on a headband device for the indications of single sided deafness or conductive hearing loss.
* Subjects will be limited to those who have no prior use of a BAI or bone conduction hearing device, normal hearing by bone conduction defined as a pure tone average of 25 dBHL or better at 500, 1000, 2000, & 3000 Hz in at least one ear. For those children where this cannot be definitively established, children will be included who display clinical signs of normal bone conduction hearing beyond a reasonable doubt and may include such evidence as (but not limited to): auditory brainstem response, speech awareness thresholds, visual reinforcement audiometry, conditioning play audiometry, CT scans, etc.)

Aim 3 a & b:

* Pediatric bilateral or unilateral conductive hearing loss patients who are between the ages of 2 and 17 years of age
* Pediatric participants who are currently managed by the University of Miami with a bone conduction device attached to a softband.

Exclusion Criteria:

Aims 1 & 2:

* Non-English speakers
* Participants reporting allergies to adhesives or highly reactive skin.

Aim 3:

* Pediatric participants who are non-English speakers.
* Children who have previous experience with a BAI or bone conduction hearing device will not be included for study.
* Pediatric participants reporting allergies to adhesives or highly reactive skin.

Aims 3a & 3b:

* Pediatric participants who are non-English speakers.
* Pediatric participants reporting allergies to adhesives or highly reactive skin.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Snapp, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Otolaryngology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adhear Followed by BAHA (Aim 3) Group: Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss or single-sided deafness who have not previously used a bone conduction device, will be provided with the Adhear system for 2 weeks (plus up to 90 days) followed by bone anchored hearing aid (BAHA) for another 2 weeks (plus up to 90 days).
  Adhear Bone Conduction System: Non-invasive bone conduction hearing device using adhesive
  Bone anchored hearing aid (BAHA): Non-invasive bone conduction hearing device using a headband
- BAHA Followed by Adhear (Aim 3) Group: Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss or single-sided deafness who have not previously used a bone conduction device, will be provided with the BAHA system for 2 weeks (plus up to 90 days) followed by Adhear for another 2 weeks (plus up to 90 days).
  Adhear Bone Conduction System: Non-invasive bone conduction hearing device using adhesive
  Bone anchored hearing aid (BAHA): Non-invasive bone conduction hearing device using a headband
Period: Overall Study
Arm/Group | Single-Sided Deafness Adult (Aim1) Group | Conductive Hearing Loss Adult (Aim 2) Group | Adhear Followed by BAHA (Aim 3) Group | BAHA Followed by Adhear (Aim 3) Group | Pediatric Unilateral Conductive Hearing Loss (Aim 3a) Group | Pediatric Bilateral Conductive Hearing Loss (Aim 3b) Group
Started | 9 | 3 | 18 | 15 (One child did not sign consent.) | 17 (Two parents consented for one child.) | 4
Received Intervention | 8 (Withdrew consent prior to receiving intervention.) | 3 | 18 | 12 (One parent child dyad screen failed. One parent consented while child did not consent, therefore, dyad screen failed.) | 14 (One of two parents of a single child participant withdrew consent. And one parent child dyad withdrew consent prior to receiving intervention.) | 4
Completed | 8 | 2 | 18 | 10 | 10 | 3
Not Completed | 1 | 1 | 0 | 5 | 7 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3 | 5 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Sided Deafness Adult (Aim1) Group | Conductive Hearing Loss Adult (Aim 2) Group | Adhear Followed by BAHA (Aim 3) Group | BAHA Followed by Adhear (Aim 3) Group | Pediatric Unilateral Conductive Hearing Loss (Aim 3a) Group | Pediatric Bilateral Conductive Hearing Loss (Aim 3b) Group | Total
Number analyzed (Participants) | 9 | 3 | 18 | 15 | 17 | 4 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 9 | 7 | 8 | 2 | 26
  Between 18 and 65 years | 8 | 3 | 9 | 8 | 9 | 2 | 39
  >=65 years | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 11 | 8 | 12 | 3 | 41
  Male | 3 | 2 | 7 | 7 | 5 | 1 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 9 | 9 | 11 | 3 | 39
  Not Hispanic or Latino | 3 | 1 | 3 | 1 | 3 | 1 | 12
  Unknown or Not Reported | 0 | 1 | 6 | 5 | 3 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 1 | 0 | 3
  White | 7 | 2 | 11 | 10 | 11 | 4 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 7 | 5 | 5 | 0 | 18

OUTCOME MEASURES:

1. Primary Outcome: Aided Hearing Thresholds for Single Sided Deafness
Description: Aided-hearing thresholds represent the softest sound that the participant can hear inside the audiometric test booth when using a hearing device. Aided hearing thresholds were measured using the participant's own device on their abutment and the Adhear device in the test booth on day 1. Hearing thresholds were measured in hertz.
Time Frame: Day 1
Population: This outcome measure corresponds to Aim 1. Overall number of participants analyzed are those participants who received the intervention and/or completed up to the visit.
Measure: Mean (Standard Deviation); unit: hertz
Groups:
- BAHA Implant: Device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant were tested with their BAHA
- Adhear Pre: Device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant were tested with the Adhear.
Arm/Group | BAHA Implant | Adhear Pre
Number analyzed (Participants) | 8 | 8
hertz
  Frequency 250 | 36.25 (7.44) | 35.63 (10.16)
  Frequency 500 | 28.13 (6.51) | 37.50 (7.07)
  Frequency 1000 | 20 (2.67) | 30.63 (6.23)
  Frequency 2000 | 23.13 (2.59) | 35.00 (8.45)
  Frequency 3000 | 27.5 (5.35) | 44.38 (4.17)
  Frequency 4000 | 33.13 (5.94) | 51.25 (6.94)
  Frequency 6000 | 31.88 (6.51) | 56.88 (5.30)
  Frequency 8000 | 40 (11.65) | 56.88 (7.53)

2. Primary Outcome: Aided Hearing Thresholds for Conductive Hearing Loss
Description: as for outcome 1
Time Frame: Day 1
Population: This outcome measure corresponds to Aim 2. Overall number of participants analyzed are those participants who received the intervention and/or completed up to the visit.
Measure: Mean (Standard Deviation); unit: hertz
Arm/Group | BAHA Implant | Adhear Pre
Number analyzed (Participants) | 3 | 3
hertz
  Frequency 250 | 17.5 (3.54) | 27.5 (3.54)
  Frequency 500 | 12.5 (10.61) | 20 (0)
  Frequency 1000 | 22.50 (3.54) | 22.5 (3.54)
  Frequency 2000 | 27.5 (3.54) | 30 (7.07)
  Frequency 3000 | 35 (0) | 40 (7.07)
  Frequency 4000 | 37.5 (10.61) | 55 (7.07)
  Frequency 6000 | 40 (14.14) | 50 (7.07)
  Frequency 8000 | 47.5 (3.54) | 55 (7.07)

3. Primary Outcome: Aided Hearing Thresholds for Single Sided Deafness
Description: Aided-hearing thresholds represent the softest sound that the participant can hear inside the audiometric test booth when using a hearing device. Aided hearing thresholds were measured using the participant's own device on a softband and the Adhear device in the test booth on day 14. Hearing thresholds were measured in hertz.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hertz
Groups:
- Baha Softband: Device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant were tested with their BAHA on softband. Placed acutely.
- Adhear Post: Device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant were tested with the Adhear system.
Arm/Group | Baha Softband | Adhear Post
Number analyzed (Participants) | 8 | 8
hertz
  Frequency 250 | 37.5 (6.78) | 31.88 (11.27)
  Frequency 500 | 31.75 (9.11) | 32.13 (9.63)
  Frequency 1000 | 24.38 (7.01) | 28.38 (4.98)
  Frequency 2000 | 28.88 (6.60) | 31.75 (7.40)
  Frequency 3000 | 35.38 (6.91) | 42.88 (4.82)
  Frequency 4000 | 45.25 (6.36) | 50.75 (7.80)
  Frequency 6000 | 46.5 (10.73) | 53.88 (7.51)
  Frequency 8000 | 50.50 (6.37) | 54.25 (7.21)

4. Primary Outcome: Aided Hearing Thresholds for Conductive Hearing Loss
Description: as for outcome 3
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hertz
Arm/Group | Baha Softband | Adhear Post
Number analyzed (Participants) | 3 | 3
hertz
  Frequency 250 | 17.5 (3.54) | 22.5 (3.54)
  Frequency 500 | 12.5 (10.61) | 25 (14.14)
  Frequency 1000 | 22.5 (3.54) | 17.5 (3.54)
  Frequency 2000 | 27.5 (3.54) | 35 (14.14)
  Frequency 3000 | 35 (0) | 47.5 (10.61)
  Frequency 4000 | 37.50 (10.61) | 55 (14.14)
  Frequency 6000 | 40 (14.14) | 50 (14.14)
  Frequency 8000 | 47.5 (3.54) | 57.5 (10.61)

5. Primary Outcome: Aided Hearing Thresholds
Description: Aided-hearing thresholds represent the softest sound that the participant can hear inside the audiometric test booth when using a hearing device. Aided hearing thresholds were measured using a traditional bone conduction device on a softband and the Adhear device in the test booth on day 14. Hearing thresholds were measured in hertz.
Time Frame: Day 14 of the intervention
Population: This outcome measure corresponds to Aim 3, Aim 3a, and Aim 3b. Overall number of participants analyzed are those participants who received the intervention and/or completed up to the visit. Insufficient sample collected for participants and thus the data could not be analyzed for arms BAHA Bilateral Conductive Hearing Loss Prior BAI Use and Adhear Bilateral Conducive Hearing Loss Prior BAI Use.
Measure: Mean (Standard Deviation); unit: hertz
Groups:
- BAHA Conductive Hearing Loss No Prior Bone Anchored Implant Use; Adhear for Conductive Hearing Loss No Prior Bone Anchored Implant Use: Pediatric participants with no prior BAI use were tested. Participant can have unilateral or bilateral conductive hearing loss.
- BAHA Unilateral Conductive Hearing Loss Prior BAI Use: Device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant were tested with a BAHA. Participant can have unilateral or bilateral conductive hearing loss.
- Adhear Unilateral Conductive Hearing Loss Prior BAI Use: Pediatric unilateral conductive hearing loss patients who are between the ages of 2 and 17 years of age with a bone conduction device attached to a softband. Subjects will be given the ADHEAR bone conduction system on trial for 2 weeks ± 90 days.
- BAHA Bilateral Conductive Hearing Loss Prior BAI Use; Adhear Bilateral Conducive Hearing Loss Prior BAI Use: Pediatric bilateral conductive hearing loss patients who are between the ages of 2 and 17 years of age with a bone conduction device attached to a softband. Subjects will be given the ADHEAR bone conduction system on trial for 4 weeks ± 7 days.
Arm/Group | BAHA Conductive Hearing Loss No Prior Bone Anchored Implant Use | Adhear for Conductive Hearing Loss No Prior Bone Anchored Implant Use | BAHA Unilateral Conductive Hearing Loss Prior BAI Use | Adhear Unilateral Conductive Hearing Loss Prior BAI Use | BAHA Bilateral Conductive Hearing Loss Prior BAI Use | Adhear Bilateral Conducive Hearing Loss Prior BAI Use
Number analyzed (Participants) | 33 | 33 | 17 | 17 | 1 | 1
hertz
  Frequency 250 | 19.43 (6.44) | 28 (9.76) | 24.17 (2.04) | 24 (7.41) | 15 (NA) — Standard Deviation not calculable for 1 participant. | 30 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 500 | 15.64 (6.54) | 24.57 (7.51) | 22.50 (5.24) | 21 (6.52) | 10 (NA) — Standard Deviation not calculable for 1 participant. | 15 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 1000 | 13.64 (7.47) | 21.43 (4.97) | 22.50 (8.22) | 22 (6.71) | 15 (NA) — Standard Deviation not calculable for 1 participant. | 20 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 2000 | 18.86 (5.17) | 24.86 (6.71) | 22.50 (4.18) | 27 (8.36) | 15 (NA) — Standard Deviation not calculable for 1 participant. | 20 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 3000 | 24.43 (6.85) | 34 (8.23) | 30 (6.32) | 28 (12.54) | 30 (NA) — Standard Deviation not calculable for 1 participant. | 40 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 4000 | 26.50 (5.81) | 39.71 (8.48) | 30 (7.07) | 32 (11.51) | 30 (NA) — Standard Deviation not calculable for 1 participant. | 35 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 6000 | 26.71 (5.30) | 37.64 (8.99) | 35 (10.48) | 37 (10.37) | 25 (NA) — Standard Deviation not calculable for 1 participant. | 30 (NA) — Standard Deviation not calculable for 1 participant.
  Frequency 8000 | 30.43 (6.52) | 37.5 (8.49) | 38.33 (17.22) | 44 (12.94) | 25 (NA) — Standard Deviation not calculable for 1 participant. | 30 (NA) — Standard Deviation not calculable for 1 participant.

6. Secondary Outcome: Aided Speech-in-noise Performance in Participants With Single-sided Deafness
Description: Aided speech-in-noise performance is the ability to identify spoken words when background noise is present while using a hearing device. Aided speech-in-noise performance was measured using the participant's own device on their abutment and the Adhear device in the test booth on day 1. Aided speech-in-noise performance was measured in decibels.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | BAHA Implant | Adhear Pre
Number analyzed (Participants) | 8 | 8
dB
  Speech front / Noise Front | 1.75 (2.46) | 1.81 (2.25)
  Speech poorer ear / Noise better ear | 2 (4.51) | 5.75 (3.87)
  Speech better ear / noise poorer ear | -2.31 (2.34) | -4.31 (1.83)

7. Secondary Outcome: Aided Speech in Noise Performance in Participants With Conductive Hearing Loss
Description: as for outcome 6
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Implant | Adhear Pre
Number analyzed (Participants) | 3 | 3
dB
  Speech front / Noise Front | 0.75 (0.35) | -0.5 (0.71)
  Speech poorer ear / Noise better ear | -3 (3.54) | -1.75 (2.47)
  Speech better ear / noise poorer ear | -6.5 (0.00) | -6.5 (1.41)

8. Secondary Outcome: Aided Speech in Noise Performance in Participants With Single-sided Deafness
Description: Aided speech-in-noise performance is the ability to identify spoken words when background noise is present while using a hearing device. Aided speech-in-noise performance was measured using the participant's own device on a softband and the Adhear device in the test booth on day 14. Aided speech-in-noise performance was measured in decibels.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Softband | Adhear Post
Number analyzed (Participants) | 8 | 8
dB
  Speech front/noise front | 0.5 (1.98) | 0.875 (1.53)
  Speech poorer ear/noise better ear | 3.81 (3.54) | 3.69 (4.29)
  Speech better ear/noise poorer ear | -4.25 (2.58) | -4.19 (2.55)

9. Secondary Outcome: Aided Speech in Noise Performance in Participants With Conductive Hearing Loss
Description: as for outcome 8
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baha Softband | Adhear Post
Number analyzed (Participants) | 3 | 3
dB
  Speech front/noise front | -1.5 (0.71) | -2.25 (1.77)
  Speech poorer ear/noise better ear | -0.5 (3.54) | -1.5 (2.83)
  Speech better ear/noise poorer ear | -7 (0.71) | -7.5 (0.00)

10. Secondary Outcome: Participant Satisfaction With BAHA (Aims 1, 2, 3a and 3b) or No Device (Aim 3)
Description: Custom Subjective Device Questionnaire measured auditory, social emotional, and device satisfaction as a composite score using a Likert scale. Likert score range was 1-4. Higher scores denoted positive responses. The reported values represent an average across the multiple domains of the questionnaire.
Time Frame: Day 1
Population: This outcome measure corresponds to Aims 1, 2, 3, 3a, and 3b. Overall number of participants analyzed are those participants who received the intervention and/or completed up to the visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baha Aim 1 Day 1: Adult participants with single-sided deafness and are experienced bone conduction device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant will be provided with the Adhear system for 2 weeks (plus up to 90 days).
- Baha Aim 2 Day 1: Adult participants with conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant will be provided with the Adhear system for 2 weeks (plus up to 90 days).
- No Device Aim 3 Day 1: Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss or single-sided deafness who have not previously used a bone conduction device, will be provided with the Adhear system for 3 weeks (plus up to 90 days) followed by bone anchored hearing aid (BAHA) for another 3 weeks (plus up to 90 days).
- Baha Subject Aim 3a Day 1: Pediatric participants (aged 2-17 years) and their parents with unilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system for 2 weeks (plus up to 90 days).
  Adhear Bone Conduction System: Non-invasive bone conduction hearing device using adhesive
- BAHA Aim 3b Day 1: Pediatric participants (aged 2-17 years) and their parents with bilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system. Participants who are fitted bilaterally will receive 2 Adhear systems (one for each ear) for 2 weeks (plus up to 90 days) at Visit 1. Participants who are fitted unilaterally will receive 1 Adhear system for 2 weeks (plus up to 90 days) at Visit 1, afterwards, will be fitted bilaterally at Visit 2 and receive the Adhear system for both ears for another 2 weeks (plus up to 90 days) for a total of 4 weeks (plus up to 180 days).
  Adhear Bone Conduction System: Non-invasive bone conduction hearing device using adhesive
Arm/Group | Baha Aim 1 Day 1 | Baha Aim 2 Day 1 | No Device Aim 3 Day 1 | Baha Subject Aim 3a Day 1 | BAHA Aim 3b Day 1
Number analyzed (Participants) | 8 | 3 | 28 | 14 | 3
score on a scale
  Subject: number analyzed (Participants) | 8 | 3 | 14 | 7 | 1
  Subject | 3.28 (0.091) | 3.88 (1.09) | 2.43 (0.52) | 2.27 (0.80) | 2.06 (1.37)
  Parent: number analyzed (Participants) | 0 | 0 | 14 | 7 | 2
  Parent |  |  | 2.55 (0.52) | 2.71 (0.51) | 3.03 (0.59)

11. Secondary Outcome: Participant Satisfaction With Adhear
Description: as for outcome 10
Time Frame: Day 14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adhear Aim 1 Day 14: Adult participants with single-sided deafness and are experienced bone conduction device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant will be provided with the Adhear system for 2 weeks (plus up to 90 days).
- Adhear Aim 2 Day 14: Adult participants with conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use and no intermittent use within the last 2 weeks) with an abutment implant will be provided with the Adhear system for 2 weeks (plus up to 90 days).
- Adhear Aim 3 Day 14: Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss or single-sided deafness who have not previously used a bone conduction device, will be provided with the Adhear system for 3 weeks (plus up to 90 days) followed by bone anchored hearing aid (BAHA) for another 3 weeks (plus up to 90 days).
- Adhear Aim 3a Day 14: Pediatric participants (aged 2-17 years) and their parents with unilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system for 2 weeks (plus up to 90 days).
- Adhear Aim 3b Day 14: Pediatric participants (aged 2-17 years) and their parents with bilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system. Participants who are fitted bilaterally will receive 2 Adhear systems (one for each ear) for 2 weeks (plus up to 90 days) at Visit 1. Participants who are fitted unilaterally will receive 1 Adhear system for 2 weeks (plus up to 90 days) at Visit 1, afterwards, will be fitted bilaterally at Visit 2 and receive the Adhear system for both ears for another 2 weeks (plus up to 90 days) for a total of 4 weeks (plus up to 180 days).
Arm/Group | Adhear Aim 1 Day 14 | Adhear Aim 2 Day 14 | Adhear Aim 3 Day 14 | Adhear Aim 3a Day 14 | Adhear Aim 3b Day 14
Number analyzed (Participants) | 8 | 3 | 28 | 14 | 3
score on a scale
  Subject: number analyzed (Participants) | 8 | 3 | 14 | 7 | 1
  Subject | 3.22 (0.86) | 3.54 (0.72) | 2.88 (0.51) | 3.38 (0.56) | 3.33 (1.20)
  Parent: number analyzed (Participants) | 0 | 0 | 14 | 7 | 2
  Parent |  |  | 2.99 (0.57) | 3.01 (0.71) | 3.24 (0.94)

12. Secondary Outcome: Participant Satisfaction With Adhear at Day 28 (Aim 3b)
Description: as for outcome 10
Time Frame: Day 28
Population: This outcome measure corresponds to Aim 3b.Overall number of participants analyzed are those participants who received the intervention and/or completed up to the visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adhear Aim 3b: Pediatric participants (aged 2-17 years) and their parents with bilateral conductive hearing loss and are experienced bone conduction device users (6 months minimum of bone conduction device use) on a headband will be provided with the Adhear system. Participants who are fitted bilaterally will receive 2 Adhear systems (one for each ear) for 2 weeks (plus up to 90 days) at Visit 1. Participants who are fitted unilaterally will receive 1 Adhear system for 2 weeks (plus up to 90 days) at Visit 1, afterwards, will be fitted bilaterally at Visit 2 and receive the Adhear system for both ears for another 2 weeks (plus up to 90 days) for a total of 4 weeks (plus up to 180 days).
  Adhear Bone Conduction System: Non-invasive bone conduction hearing device using adhesive
Arm/Group | Adhear Aim 3b
Number analyzed (Participants) | 3
score on a scale
  Subject: number analyzed (Participants) | 1
  Subject | 2.87 (0.48)
  Parent: number analyzed (Participants) | 2
  Parent | 2.94 (0.49)

ADVERSE EVENTS:
Time Frame: 506 days
Groups:
- Adhear (Aim 3) Group: Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss who have not previously used a bone conduction device, will be provided with the Adhear system for 2 weeks (plus up to 90 days).
  Adhear Bone Conduction System: Non-invasive bone conduction hearing device using adhesive
- BAHA (Aim 3) Group: Pediatric participants (aged 5-17 years) and their parents with conductive hearing loss who have not previously used a bone conduction device, will be provided with the BAHA system for 2 weeks (plus up to 90 days).
  Bone anchored hearing aid (BAHA): Non-invasive bone conduction hearing device using a headband
Arm/Group | Single-Sided Deafness Adult (Aim1) Group | Conductive Hearing Loss Adult (Aim 2) Group | Adhear (Aim 3) Group | BAHA (Aim 3) Group | Pediatric Unilateral Conductive Hearing Loss (Aim 3a) Group | Pediatric Bilateral Conductive Hearing Loss (Aim 3b) Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/33 | 0/33 | 0/14 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/33 | 0/33 | 0/14 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/33 | 0/33 | 0/14 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03533686/Prot_SAP_000.pdf